CLINICAL TRIAL: NCT04358783
Title: Phase II, Randomized, Double-blind, Controlled Clinical Trial Evaluating the Efficacy and Safety of Plasma From Patients Cured of COVID-19 Compared to the Best Available Therapy in Subjects With SARS-CoV-2 Pneumonia
Brief Title: Convalescent Plasma Compared to the Best Available Therapy for the Treatment of SARS-CoV-2 Pneumonia
Acronym: COP-COVID-19
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hospital Universitario Dr. Jose E. Gonzalez (Other)
Responsible Party: Principal Investigator, Dr. Adrian Camacho-Ortiz, Head of the Infectious Disease Department, Hospital Universitario Dr. Jose E. Gonzalez
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IF20-00002
Record Dates: First submitted 2020-04-21; First posted 2020-04-24 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: Coronavirus Infection
Keywords: COVID-19; Plasma from patients cured; SARS-CoV-2 pneumonia
MeSH Terms: conditions — Coronavirus Infections; COVID-19

STUDY DESIGN:
Intervention Model Description: RCT double blind comparative study
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: double blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Plasma (Experimental): Convalescent plasma from cured COVID-19 patients y Supportive management depending on individual needs
  Interventions: Biological: Plasma
- Best Available Therapy (Experimental): Will receive supportive management depending on individual needs including.
  Interventions: Other: Best Available Therapy

INTERVENTIONS:
Biological: Plasma — The plasma unit will be fractionated in 200 mL aliquots for storage at -80°C until use. After thawing, it shall be administered in a single 200 mL dose to subjects who are randomized to that arm.
  Arms: Plasma
Other: Best Available Therapy — It shall include, but not be limited to, oxygen therapy by means of a nasal cannula; high-flow nasal cannula; invasive or non-invasive mechanical ventilation; intravenous hydration; antibiotic therapy; thrombus prophylaxis; pain and fever management.
  Arms: Best Available Therapy

SUMMARY:
In early December 2019, cases of pneumonia of unknown origin were identified in Wuhan, China. The causative virus was called severe acute respiratory syndrome coronavirus 2 (SARS-CoV-2). The World Health Organization (WHO) has recently declared coronavirus disease 2019 (COVID-19) a public health emergency of international concern.

According to the World Health Organization (WHO), the management of COVID-19 has focused primarily on infection prevention, detection and patient monitoring. However, there is no vaccine or specific treatment for SARS-CoV-2 due to the lack of evidence. Treatment options currently include broad-spectrum antiviral drugs but the efficacy and safety of these drugs is still unknown.

Convalescent plasma has previously been used to treat various outbreaks of other respiratory infections; however, it has not been shown to be effective in all the diseases studied. Therefore, clinical trials are required to demonstrate its safety and efficacy in patients with VIDOC-19.

The present work seeks to determine the mortality from any cause up to 14 days after plasma randomization of patients cured of COVID-19 compared to the Best Available Therapy in subjects with SARS-CoV-2 pneumonia. This is a 2:1 randomized, double-blind, single-center, phase 2, controlled clinical trial (plasma: best available therapy) for the treatment of SARS-CoV-2 pneumonia.

DETAILED DESCRIPTION:
Randomized clinical trial comparing convalescent plasma to best available therapy (BAT) for the treatment of severely ill and critically ill patient with COVID-19: Patients will be electronically randomized 2:1 (plasma vs BAT) in a double blind fashion. Patients with SARS-CoV-2 PCR confirmed infection with pulmonary infiltrates and hypoxemia will be screened and invited to participate. Primary outcomes will be early all-cause mortality, and secondary outcomes will include all cause in hospital mortality, length of mechanical ventilation and hospital stay, time to PAO2 >200, progression of pulmonary infiltrates, antibody titers and time to negative PCR detection

ELIGIBILITY:
Inclusion Criteria:

1. Men or women ≥18 years. If you are a woman of childbearing age, you must agree to practice abstinence or to use an effective method of contraception during the study period.
2. Vascular access suitable for administration of hemocomponents.
3. SARS-CoV-2 positive RT-PCR.
4. Negative pregnancy test in case of a woman of reproductive age
5. Signing of evidentiary document of informed consent.
6. Hospital admission for SARS-CoV-2 pneumonia with supplemental oxygen requirements.
7. Subjects who access the storage of biological samples for future examination.

Exclusion Criteria:

1. Respiratory rate >30 RPM, SO2 <93%, PaO2/FiO2 <200 despite intervention with oxygen therapy after 60 minutes of hospitalization.
2. New alteration of the state of alert that does not revert after interventions 60 minutes after admission to hospital.
3. PAM ≤ 65mmHg despite initial resuscitation on arrival at the centre.
4. Pregnant or breastfeeding patients.
5. Patients that the investigators consider inappropriate to participate in the clinical trial
6. Contraindication to transfusion or history of previous severe reaction to blood products.
7. Have received any blood products in the last 120 days.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-04-27 (Actual); Primary Completion 2021-05-01 (Actual); Study Completion 2021-05-01 (Actual)

PRIMARY OUTCOMES:
Early all-cause mortality | 14 days
  any cause mortality during the first 14 days of treatment

SECONDARY OUTCOMES:
Time in days for SARS-CoV-2 RT-PCR negatives | 90 days
  (48-hour sampling interval from day 3 of hospitalization to two consecutive negatives).
The serum anti-SARS-CoV-2 antibody titres | 90 days
  In subjects of both arms at day 0, 3, 7, 14 and 90.
Detection of serum antibodies | days 0, 3, 7, 14 and 90.
  Comparison of anti-SARS-CoV-2 antibody titers

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Camacho-Ortiz, MD, Principal Investigator — Hospital Universitario "Dr. Jose Eleuterio Gonzalez, UANL
Locations (1):
- Hospital Universitario José E. Gonzalez, Monterrey, Nuevo León, Mexico

REFERENCES:
- [Background] Guan WJ, Ni ZY, Hu Y, Liang WH, Ou CQ, He JX, Liu L, Shan H, Lei CL, Hui DSC, Du B, Li LJ, Zeng G, Yuen KY, Chen RC, Tang CL, Wang T, Chen PY, Xiang J, Li SY, Wang JL, Liang ZJ, Peng YX, Wei L, Liu Y, Hu YH, Peng P, Wang JM, Liu JY, Chen Z, Li G, Zheng ZJ, Qiu SQ, Luo J, Ye CJ, Zhu SY, Zhong NS; China Medical Treatment Expert Group for Covid-19. Clinical Characteristics of Coronavirus Disease 2019 in China. N Engl J Med. 2020 Apr 30;382(18):1708-1720. doi: 10.1056/NEJMoa2002032. Epub 2020 Feb 28. PMID 32109013
- [Background] Rothan HA, Byrareddy SN. The epidemiology and pathogenesis of coronavirus disease (COVID-19) outbreak. J Autoimmun. 2020 May;109:102433. doi: 10.1016/j.jaut.2020.102433. Epub 2020 Feb 26. PMID 32113704
- [Background] Zhang L, Liu Y. Potential interventions for novel coronavirus in China: A systematic review. J Med Virol. 2020 May;92(5):479-490. doi: 10.1002/jmv.25707. Epub 2020 Mar 3. PMID 32052466
- [Background] Wu Z, McGoogan JM. Characteristics of and Important Lessons From the Coronavirus Disease 2019 (COVID-19) Outbreak in China: Summary of a Report of 72 314 Cases From the Chinese Center for Disease Control and Prevention. JAMA. 2020 Apr 7;323(13):1239-1242. doi: 10.1001/jama.2020.2648. No abstract available. PMID 32091533
- [Background] Numbers SIN. Coronavirus Disease 2019 ( COVID-19 ) Situation Report-71. Vol 2019.; 2020.
- [Background] Heymann DL, Shindo N; WHO Scientific and Technical Advisory Group for Infectious Hazards. COVID-19: what is next for public health? Lancet. 2020 Feb 22;395(10224):542-545. doi: 10.1016/S0140-6736(20)30374-3. Epub 2020 Feb 13. No abstract available. PMID 32061313
- [Background] Disease C. Interim Clinical Guidance for Management of Patients with Confirmed Coronavirus Disease ( COVID-19 ). CDC. 2020;2019:4-6.
- [Background] Yang Y, Yang M, Shen C, Wang F, Yuan J. Evaluating the accuracy of different respiratory specimens in the laboratory diagnosis and monitoring the viral shedding of 2019-nCoV infections ABSTRACT : medRxiv. 2020.
- [Background] Guidance I. Clinical management of severe acute respiratory infection ( SARI ) when COVID-19 disease is suspected . World Heal Organ. 2020:1-21.
- [Background] Lu H. Drug treatment options for the 2019-new coronavirus (2019-nCoV). Biosci Trends. 2020 Mar 16;14(1):69-71. doi: 10.5582/bst.2020.01020. Epub 2020 Jan 28. PMID 31996494
- [Background] Casadevall A, Pirofski LA. The convalescent sera option for containing COVID-19. J Clin Invest. 2020 Apr 1;130(4):1545-1548. doi: 10.1172/JCI138003. No abstract available. PMID 32167489
- [Background] Cheng Y, Wong R, Soo YO, Wong WS, Lee CK, Ng MH, Chan P, Wong KC, Leung CB, Cheng G. Use of convalescent plasma therapy in SARS patients in Hong Kong. Eur J Clin Microbiol Infect Dis. 2005 Jan;24(1):44-6. doi: 10.1007/s10096-004-1271-9. PMID 15616839
- [Background] Hung IF, To KK, Lee CK, Lee KL, Chan K, Yan WW, Liu R, Watt CL, Chan WM, Lai KY, Koo CK, Buckley T, Chow FL, Wong KK, Chan HS, Ching CK, Tang BS, Lau CC, Li IW, Liu SH, Chan KH, Lin CK, Yuen KY. Convalescent plasma treatment reduced mortality in patients with severe pandemic influenza A (H1N1) 2009 virus infection. Clin Infect Dis. 2011 Feb 15;52(4):447-56. doi: 10.1093/cid/ciq106. Epub 2011 Jan 19. PMID 21248066
- [Background] Sahr F, Ansumana R, Massaquoi TA, Idriss BR, Sesay FR, Lamin JM, Baker S, Nicol S, Conton B, Johnson W, Abiri OT, Kargbo O, Kamara P, Goba A, Russell JB, Gevao SM. Evaluation of convalescent whole blood for treating Ebola Virus Disease in Freetown, Sierra Leone. J Infect. 2017 Mar;74(3):302-309. doi: 10.1016/j.jinf.2016.11.009. Epub 2016 Nov 17. PMID 27867062
- [Background] Mair-Jenkins J, Saavedra-Campos M, Baillie JK, Cleary P, Khaw FM, Lim WS, Makki S, Rooney KD, Nguyen-Van-Tam JS, Beck CR; Convalescent Plasma Study Group. The effectiveness of convalescent plasma and hyperimmune immunoglobulin for the treatment of severe acute respiratory infections of viral etiology: a systematic review and exploratory meta-analysis. J Infect Dis. 2015 Jan 1;211(1):80-90. doi: 10.1093/infdis/jiu396. Epub 2014 Jul 16. PMID 25030060
- [Background] Marano G, Vaglio S, Pupella S, Facco G, Catalano L, Liumbruno GM, Grazzini G. Convalescent plasma: new evidence for an old therapeutic tool? Blood Transfus. 2016 Mar;14(2):152-7. doi: 10.2450/2015.0131-15. Epub 2015 Nov 6. PMID 26674811
- [Background] Brunk D. FDA OKs Emergency Use of Convalescent Plasma for Seriously Ill COVID-19 Patients. medscape. 2020:28-29. doi:10.1001/jama.2020.4783
- [Background] Tanne JH. Covid-19: FDA approves use of convalescent plasma to treat critically ill patients. BMJ. 2020 Mar 26;368:m1256. doi: 10.1136/bmj.m1256. No abstract available. PMID 32217555
- [Background] Shen C, Wang Z, Zhao F, Yang Y, Li J, Yuan J, Wang F, Li D, Yang M, Xing L, Wei J, Xiao H, Yang Y, Qu J, Qing L, Chen L, Xu Z, Peng L, Li Y, Zheng H, Chen F, Huang K, Jiang Y, Liu D, Zhang Z, Liu Y, Liu L. Treatment of 5 Critically Ill Patients With COVID-19 With Convalescent Plasma. JAMA. 2020 Apr 28;323(16):1582-1589. doi: 10.1001/jama.2020.4783. PMID 32219428
- [Background] Roback JD, Guarner J. Convalescent Plasma to Treat COVID-19: Possibilities and Challenges. JAMA. 2020 Apr 28;323(16):1561-1562. doi: 10.1001/jama.2020.4940. No abstract available. PMID 32219429
- [Background] NORMA Oficial Mexicana NOM-253-SSA1-2012, Para la disposición de sangre humana y sus componentes con fines terapéuticos. D Of. 2012;Tercera Se.